CLINICAL TRIAL: NCT04415502
Title: CTHRC1: A Biomarker for Evaluation of Rheumatoid Arthritis Disease Activity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lobna Amer Araby Ahmed, Principal investigator, Assiut University
Other Study IDs: CTHRC1 in RA
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Measuring of CTHRc1 , its correlation with RAdisease activity: Measuring of CTHRc1 levels and its correlation with RA disease activity

SUMMARY:
The purpose of the study is to determine whether plasma levels of the collagen triple helix repeat containing (CTHRC1) protein can serve as a blood-based biomarker for diagnosis of rheumatoid arthritis (RA) ,and furthermore its correlation with disease activity

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, progressive, autoimmune disease of synovial joints. Characterized by periods of flares with high disease activity involving both a systemic immune response and tissue-specific inflammatory events that can lead to erosive joint and bone destruction and subsequent disability . Currently, diagnosis of RA is based mainly on the extent of tenderness and swelling of the joints , levels of acute-phase reactants such as C-reactive protein (CRP) ,erythrocyte sedimentation rate(ESR) , high titers of rheumatoid factor (RF) and high titers of antibodies against cyclic citrullinated peptide (anti-CCP) in the plasma .Recently, reported increased levels of collagen triple helix repeat containing 1 protein (CTHRC1) are strongly associated with the severity of murine proteoglycan-induced arthritis and collagen antibody-induced murine arthritis (CAIA) , further CTHRC1 expression in murine experimental arthritis is increased in the synovium and specifically detected in activated murine , located at the synovial intimal lining and at the bone-pannus interface .Of interest,The expression pattern of CTHRC1 in pannus, its role in the function of FLS relevant to cartilage damage in RA, and CTHRC1's association with disease severity in murine arthritis raised the question of whether CTHRC1 could be used as a marker for RA diagnosis and monitoring of disease activity in patients .

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as RA
* age more than 18 years

Exclusion Criteria:

* other rheumatological diseases Malignancies Hepatic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Measuring of CTHRc1 levels and its correlation with RA disease activity
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
CTHRC1 in RA | One year
  Measuring of CTHRc1 in Rheumatoid arthritis patients.
CTHRc1 and RA disease activity | One year
  Correlation of CTHRc1levels with RA disease activity

REFERENCES:
- [Background] Chewick S. Infection control demand administrative support. Dimens Health Serv. 1975 Dec;52(12):40-1. No abstract available. PMID 1305
- [Background] Lumholtz IB. [Nurses' drug information: therapeutic action group: benzodiazepine derivatives. 2]. Sygeplejersken. 1975 Sep 24;75(38):15. No abstract available. Danish. PMID 803